CLINICAL TRIAL: NCT04501068
Title: Analysis of 150 Consecutive Uses of the Ambu® AuraGain Supraglottic Airway by One Anaesthetist in Ambulatory Surgery
Brief Title: Evaluation of the Ambu® AuraGain in Ambulatory Surgery
Status: Completed | Type: Observational
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Matilde Zaballos, Anesthesiologist, Hospital General Universitario Gregorio Marañon
Other Study IDs: MULTIAURAGAIN
Record Dates: First submitted 2020-07-28; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Airway
Keywords: Ambu® AuraGainTM; Second Generation Laryngeal Masks Airway

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ambu AuraGain: Ambu® AuraGainTM Patients undergoing anesthesia in which airway management includes a Ambu® AuraGainTM supraglottic airway and fulfill the inclusion criteria of the study.
  Interventions: Device: Ambu® AuraGainTM

INTERVENTIONS:
Device: Ambu® AuraGainTM — Evaluate the time of insertion, performance, security and insertion success rate of the Ambu® AuraGainTM in patients undergoing ambulatory surgery and general anaesthesia

SUMMARY:
The study was designed to evaluate the success rate, time of insertion, sealing efficacy and security of the Ambu® AuraGain in patients undergoing ambulatory surgery by one anesthetist

DETAILED DESCRIPTION:
Supraglottic devices (SGD), in all their different forms, have become an authentic innovation in airway management especially in day surgery. The Ambu® AuraGainTM (Ambu A/S, Ballerup, Denmark) is a new single-use, anatomically curved supraglottic airway with an integrated gastric access port designed to provide functional separation of the respiratory and digestive tracts allowing the exit of gastric contents and the passage of a gastric tube to manage gastric contents.

Its characteristics in the design, composition by a smooth and atraumatic material, the presence of the gastric drainage access, with potential improved patient safety and its characteristic of being disposable, suggests a significant expansion of its use in the coming years.

The series in the literature reporting performance or safety of use of the Ambu® AuraGainTM come from studies on selected cases and in certain surgical procedures. However, there are limited studies that have evaluated the efficacy of the device in routine clinical practice in patients intervened in ambulatory surgery and performed by a single investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery procedures in ambulatory surgery usually performed with supraglottic devices.
* ASA physical status I-III patients
* Age 18-no limit

Exclusion Criteria:

* Patients with known difficult airway
* Patients with increased risk of aspiration
* Patient refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for outpatient surgery. Patients who require the insertion of a supraglottic device as part of their anesthetic management.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the number of attempts to insert the Ambu® AuraGainTM supraglottic airway | The number of insertion attempts will be collected after anesthesia induction
  Insertion attempts (in numbers)
  From picking up the Ambu® AuraGainTM supraglottic airway until the mask is placed into the patient mouth. (in numbers)
Evaluate the time to insert the Ambu® AuraGainTM supraglottic airway | The insertion time will be collected after anesthesia induction after administration of propofol
  The time from picking up the Ambu® AuraGainTM supraglottic airway until the cuff was inflated. (in seconds)

SECONDARY OUTCOMES:
Blood pressure during insertion of the Ambu® AuraGainTM supraglottic airway | At baseline and every 3 minutes until 6 minutes after insertion of the Ambu® AuraGainTM supraglottic airway
  Blood pressure in mmHg
Heart rate during insertion of the Ambu® AuraGainTM supraglottic airway heart rate | At baseline and every 3 minutes until 6 minutes after insertion of the Ambu® AuraGainTM supraglottic airway]
  Heart rate in beep per minute
BIS data | At baseline and every 3 minutes until 6 minutes after insertion of the Ambu® AuraGainTM supraglottic airway (To evaluate the evolution of BIS values during insertion of the Ambu® AuraGainTM supraglottic airway
  Bis data: number from 100 (awake) to 40-45 (anesthetic status)
Oropharyngeal leak pressure of the Ambu® AuraGainTM supraglottic airway. | The Oropharyngeal leak pressure of the Ambu® AuraGainTM supraglottic airway will be collected 10 minutes after the Ambu® AuraGainTM supraglottic airway will be inserted]
  The Oropharyngeal leak pressure of the Ambu® AuraGainTM supraglottic airway will be determined with an intracuff pressure of 60 cm H2O by closing the expiratory valve of the breathing circle circuit at a fixed gas flow of 3 L/min and noting the pressure at which an oropharyngeal leak occurs. (in cm H2O)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Hortal, MD, PhD, Study Chair — Servicio de Anestesiología, Hospital General Universitario Gregorio Marañón
Locations (2):
- Spain (2):
  - Hospital Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Gregorio Maranon, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shariffuddin II, Teoh WH, Tang E, Hashim N, Loh PS. Ambu(R) AuraGain versus LMA Supreme Second Seal: a randomised controlled trial comparing oropharyngeal leak pressures and gastric drain functionality in spontaneously breathing patients. Anaesth Intensive Care. 2017 Mar;45(2):244-250. doi: 10.1177/0310057X1704500215. PMID 28267947
- [Result] Wong DT, Ooi A, Singh KP, Dallaire A, Meliana V, Lau J, Chung F, Singh M, Wong J. Comparison of oropharyngeal leak pressure between the Ambu(R) AuraGain and the LMA(R) Supreme supraglottic airways: a randomized-controlled trial. Can J Anaesth. 2018 Jul;65(7):797-805. doi: 10.1007/s12630-018-1120-4. Epub 2018 Mar 26. PMID 29582360
- [Result] Lopez AM, Agusti M, Gambus P, Pons M, Anglada T, Valero R. A randomized comparison of the Ambu AuraGain versus the LMA supreme in patients undergoing gynaecologic laparoscopic surgery. J Clin Monit Comput. 2017 Dec;31(6):1255-1262. doi: 10.1007/s10877-016-9963-0. Epub 2016 Nov 26. PMID 27889843
- [Result] Preece G, Ng I, Lee K, Mezzavia P, Krieser R, Williams DL, Stewart O, Segal R. A randomised controlled trial comparing fibreoptic-guided tracheal intubation through two supraglottic devices: Ambu(R) AuraGain laryngeal mask and LMA(R) Fastrach. Anaesth Intensive Care. 2018 Sep;46(5):474-479. doi: 10.1177/0310057X1804600508. PMID 30189821